CLINICAL TRIAL: NCT02265471
Title: Knowledge and Perception of Resistance to Antimicrobials in French Healthcare Facilities
Brief Title: Knowledge and Perception of Resistance to Antimicrobials Among Healthcare Workers in France
Acronym: PerceptR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PHRQ1277
Record Dates: First submitted 2014-05-27; First posted 2014-10-16 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2014-04

CONDITIONS: Knowledge, Perception and Behaviour of Resistance to Antimicrobial Among HCW

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- university hospital: university hospital
- large or small public hospitals: large or small public hospitals
- private HCFs: private HCFs
- referral centers for cancer: referral centers for cancer
- chirurgical facilities, clinic: chirurgical facilities, clinic
- mixed group: local hospitals, long term care and post-op and rehabilitation facilities, and nursing homes

SUMMARY:
The objectives of this survey are to determine the level of antimicrobial resistance knowledge and perception of health care workers (HCW) in France, to measure the impact of health care facilities (HCF) and to identify the drivers and barriers to change. To achieve this goal, a cross-sectional survey on one day with a self-administered questionnaire and semi-structured interviews with HCWs is proposed. This study will be planned in 60 different HCFs randomly selected and expected to include of 2,100 to 10,000 respondents.

DETAILED DESCRIPTION:
BACKGROUND The landscape of antibiotic resistance in hospital has dramatically evolved over the past 10 years, with rapid change of multidrug resistant organisms (MDROs), i.e. decreasing rate of methicillin-resistant Staphylococcus aureus (MRSA) and increasing prevalence of Extended-spectrum beta-lactamase (ESBL) - producing Enterobacteriaceae in the community and the hospital, emergence of highly resistant bacteria (HRB) especially vancomycin-resistant enterococci (VRE) and carbapenemase-producing Enterobacteriaceae (CPE) that are most often imported for foreign countries.

Schematically, the control of bacterial resistance is based on the modulation of antibiotics prescription and on the interruption of HRB or MDRO cross-transmission. Many recommendations have recently been issued for the management of patients carrying HRB or MDRO, but their level of knowledge and implementation in health care facilities (HCF) remains unclear.

Knowledge and perception of resistance to antimicrobials in among health care workers (HCW) are influenced by individual and societal determinants, professional environment and personal experience. The willing of improving antimicrobial resistance awareness and changing behaviors requires an accurate overview of the knowledge and perceptions of the HCW within the French health care settings.

OBJECTIVES The main objective is to determine the level of antimicrobial resistance knowledge among HCWs in France.

The secondary objectives are: 1) to determine the antimicrobial resistance perception of HCW in France; 2) to measure the impact of HCF organisation and the perception on the knowledge of HCW; 3) to identify and analyse the drivers and barriers to change.

MATERIALS AND METHODS The methodology used is a cross-sectional survey on one day with a self-administered questionnaire and semi-structured interviews with HCW (doctors, nurses and aides, employed or in training, and directly participating in care). This survey will be implemented in a random sample representative of the French HCFs. The questionnaires include data on HCF and individual data on respondents and evaluations regarding: the knowledge of HCW (landscape of resistance, the role and control of cross-transmission, the role of selective pressure caused by antibiotics), the perception of antimicrobial resistance (using the Health Belief Model), a measure of organization's workplace culture (based on leadership, commitment, team communication and level of stress / chaos). Semi-structured interviews have been planned to complement the assessment.

JUDGING CRITERIA The main criterion is the level of knowledge with binary encoding. The secondary criteria are based on the psycho-social-cognitive determinants of knowledge and perceptions and the culture of the organisation.

INCLUSIONS Six types of HCF (university hospital, large or small public hospitals, private HCFs, referral centers for cancer, and a mixed group of local hospitals, long term care and post-op and rehabilitation facilities, and nursing homes in each of the 5 interregional coordination centers for infection control (CCLIN). All eligible HCWs working during the survey day will be included. A minimum of 2,100 HCW is required to properly estimate the rate of HCW with the minimum core of knowledge (p<0.05). Actually, a larger number of 5,000 to 10,000 participants should be included.

All HCWs, employed or training, working during the day of the survey (day and night) in the selected HCF will be included except the health workers who are not involved in direct care, non-medical staff other than nurses or nursing auxiliary.

ELIGIBILITY:
Inclusion Criteria:

* doctors, nurses and aides, employed or in training, and directly participating in care

Exclusion Criteria:

* physicians not participating in care, pharmacist, laboratory employees, administrative employees

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: health care workers (medical or not)
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
percentage of healthcare workers with appropriate knowledge and related environmental conditions | 1 day
  psycho-social-cognitive determinants of knowledge and perceptions and the culture of the organisation

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe Lucet, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vaillant L, Birgand G, Esposito-Farese M, Astagneau P, Pulcini C, Robert J, Zahar JR, Sales-Wuillemin E, Tubach F, Lucet JC; PerceptR Study group. Awareness among French healthcare workers of the transmission of multidrug resistant organisms: a large cross-sectional survey. Antimicrob Resist Infect Control. 2019 Nov 12;8:173. doi: 10.1186/s13756-019-0625-0. eCollection 2019. PMID 31749961